CLINICAL TRIAL: NCT03990506
Title: Comparison of Epi-off and Epi-on Photorefractive Intrastromal Crosslinking (PiXL) for Progressive Keratoconus
Brief Title: Photorefractive Intrastromal Crosslinking (PiXL) for the Treatment of Progressive Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Glaukos Corporation (Industry)
Responsible Party: Principal Investigator, Anders Behndig, Principal Investigator, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PiXLKC-I
Record Dates: First submitted 2019-06-12; First posted 2019-06-19 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Keratoconus; Corneal Crosslinking; Corneal Biomechanics; Corneal Densitometry; Scheimpflug Photography; Corneal Disease; Eye Diseases
MeSH Terms: conditions — Keratoconus; Corneal Diseases; Eye Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, single-masked intraindividually comparing randomized controlled trial. Participants will be randomized to receive Epi-off PiXL in one eye and Epi-on PiXL in the other, which is masked to the participant. The participant can choose to treat in eye at a time or both eyes during the same visit.
Who Masked: Participant
Masking Description: The participants are not aware which eye will receive the Epi-off PiXL treatment and which eye will receive the Epi-on PiXL treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epi-on PiXL (Experimental): Photorefractive intrastromal corneal crosslinking without epithelium debridement during humidified high oxygen flow.
  Interventions: Procedure: Epi-on PiXL
- Epi-off PiXL (Active Comparator): Photorefractive intrastromal corneal crosslinking with epithelium debridement.
  Interventions: Procedure: Epi-Off PiXL

INTERVENTIONS:
Procedure: Epi-on PiXL — Photorefractive intrastromal crosslinking (PiXL) After local anaesthetics, the cornea is soaked in Riboflavin by repeated topical application during 10 minutes. For masking purposes, epithelial debridement is simulated by moving a scraping instrument in front of the cornea. A Riboflavin soaked sponge is used to lightly disrupt the epithelium tight junctions, without epithelium debridement. The cornea is illuminated with PiXL under 16:40 minutes during continuously delivery of humidified high oxygen via specific oxygen goggles. The UV-dosage is individually customized based upon Kmax; < 45D, 7.2J/cm2; 45-50D, 10J/cm2; > 50D, 15 J/cm2.
  Arms: Epi-on PiXL
Procedure: Epi-Off PiXL — Photorefractive intrastromal crosslinking (PiXL) After local anaesthetics, the corneal epithelium is debrided and the cornea is soaked in Riboflavin by repeated topical application during 10 minutes. The cornea is then illuminated with individually customized topography-guided PiXL under 16:40 minutes. The UV-dosage is individually customized based upon Kmax; < 45D, 7.2J/cm2; 45-50D, 10J/cm2; > 50D, 15 J/cm2.
  Arms: Epi-off PiXL

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and postoperative ocular discomfort by comparing individually customized Photorefractive intrastromal crosslinking (PiXL) for progressive Keratoconus. The study compares two different protocols, PiXL with corneal epithelium debridement (Epi-off) and PiXL without epithelium debridement in high oxygen environment (Epi-on), with the hypothesis that Epi-on gives less postoperative ocular discomfort.

DETAILED DESCRIPTION:
The study is designed as a prospective, single-masked intraindividually comparing randomized clinical trial involving participants of both genders aged 18-35 years with Keratoconus planned for routine corneal crosslinking at the Department of Ophthalmology, Umeå University Hospital, Umeå, Sweden. The study includes 32 participants with bilateral Keratoconus, receiving Epi-off PiXL (n=32) in one eye and Epi-on PiXL in high oxygen environment (n=32) in the fellow eye. The participants are randomized to epi-on PiXL utilizing block randomization with a sample size of 16 in each block; 16 right eyes and 16 left eyes. All participants are informed about the procedures before consenting to participate in the study.

At baseline, before treatment, each eye is examined with slit-lamp microscopy, subjective refraction, determination of uncorrected (UCVA), low contrast visual acuity at 2.5 percentage contrast and 10 percentage contrast and best corrected (BSCVA) visual acuities using the LogMAR fast protocol and intraocular pressure (IOP) using Goldmann applanation tonometry. Under standardized, mesopic light conditions each eye is evaluated by keratometry readings and central corneal thickness using Schemipflug camera measurements, Pentacam HR® (Oculus, Inc. Lynnwood, WA).

Endothelial cellcount is assessed (SP-2000P, Topcon, Inc) and total ocular wavefront is measured with iTrace (Tracey Technologies, Inc.).

Ocular discomfort is subjectively evaluated in each eye by a specific visual analogous rating scale at 4h, 8h 24h and thereafter daily up to 1 week postoperatively.

All the above mentioned examinations are repeated at 1, 3, 6, 12 and 24 months after treatment. At 1 day and 1 week after treatment, solely UCVA, Auto-refractor measurements and slit-lamp examination are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for corneal crosslinking.
* Progressive keratoconus documented with a consistent decrease of best corrected visual acuity with no other explanation, an unquestionable historical progression, or a progression documented with the Pentacam Scheimpflug camera with at least 2 of the following: progressive anterior and/or posterior corneal steepening and/or progressive corneal thinning and/or increased rate of corneal thickness change from the periphery to the center.
* A keratoconus diagnosis based on abnormal posterior elevation, abnormal corneal thickness distribution and clinical noninflammatory corneal thinning using the "Belin/Ambrósio enhanced ectasia" measurements of the Pentacam Scheimpflug camera.
* Minimum corneal thickness of 400 µm at the thinnest point before epithelial removal.
* 18-35 years of age
* No ocular abnormalities except keratoconus
* No previous ocular surgery
* No cognitive insufficiency interfering with the informed consent.

Exclusion Criteria:

* Age under 18 or over 35
* Any corneal abnormalities except keratoconus
* Pregnancy or lactation
* Previous ocular surgery
* Cognitive insufficiency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Maximal keratometry (Kmax) | 1 month, 3 months, 6 months, 12 months and 24 months after treatment
  Kmax assessed with the Pentacam HR Scheimpflug camera, Diopters.

SECONDARY OUTCOMES:
Uncorrected distance visual acuity (UDVA) | 1 month, 3 months, 6 months, 12 months and 24 months after treatment
  Change from baseline in distance uncorrected visual acuity, LogMAR
Best corrected visual acuity (BCVA) | 1 month, 3 months, 6 months, 12 months and 24 months after treatment
  Change from baseline in distance best corrected visual acuity, LogMAR
Mean keratometry (Kmean) | 1 month, 3 months, 6 months, 12 months and 24 months after treatment
  Kmean (average) assessed with the Pentacam HR Scheimpflug camera, Diopters.
Subjective Ocular Discomfort Scores | 4 hours, 8 hours, 1 day, 2 days, 3 days, 4 days, 5 days, 6 days and 7 days after treatment
  Subjective Ocular Discomfort Scores, Visual Analog Score (0 (no discomfort) - 10 (maximum discomfort)) for each eye, mm.
Low contrast visual acuity (LCVA) | 1 month, 3 months, 6 months, 12 months and 24 months after treatment
  Change from baseline in low contrast visual acuities at 10 % and 2.5 % contrast, LogMAR
Manifest spherical equivalent (MRSE) | 1 month, 3 months, 6 months, 12 months and 24 months after treatment
  Change from baseline in spherical equivalent on subjective distance refraction, Diopters
Central corneal thickness (CCT) | 1 month, 3 months, 6 months, 12 months and 24 months after treatment
  Change from baseline in central corneal thickness assessed with Pentacam, Scheimpflug camera, μm.
Change from baseline in ocular wavefront aberrometry | 1 month, 3 months, 6 months, 12 months and 24 months after treatment
  Change from baseline in higher order aberrations assessed with iTrace, Root mean square.
Endothelial cell density (ECC) | 24 months after treatment
  Change from baseline in endothelial cell density, cells/mm2
Intraocular pressure (IOP) | 1 month, 3 months, 6 months, 12 months and 24 months after treatment
  Change from baseline in intraocular pressure assessed with Goldmann applanation tonometry, mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Behndig, MD, PhD, Principal Investigator — Department of Clinical Sciences/Ophthalmology, Umeå University
Locations (1):
- Department of Clinical Sciences/Ophthalmology, Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No